CLINICAL TRIAL: NCT00522041
Title: A Randomized. Double-blind, Placebo-controlled, Multi-national Study to Determine the Effect of Cellegesic Nitroglycerin Ointment 0.4% (Cellegesic) on the Pain Associated With a Chronic Anal Fissure
Brief Title: A Study to Determine the Effect of Nitroglycerin Ointment 0.4% (Cellegesic) on the Pain Associated With Chronic Anal Fissures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-C-01
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Fissure in Ano; Pain
Keywords: Pain associated with chronic anal fissure
MeSH Terms: conditions — Fissure in Ano; Pain | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellegesic (nitroglycerin 0.4%) (Experimental): Participants applied Cellegesic 375 mg ointment containing approximately 1.5 mg of nitroglycerin anally twice daily for 21 days. In addition, participants took acetaminophen 650 mg orally twice daily for 21 days.
  Interventions: Drug: Cellegesic
- Placebo 375 mg (Placebo Comparator): Participants applied placebo 375 mg ointment anally twice daily for 21 days. In addition, participants took acetaminophen 650 mg orally twice daily for 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cellegesic — Cellegesic was supplied as an ointment containing 0.4% w/w nitroglycerin.
  Other Names: 0.4% nitroglycerin ointment; Rectogesic
  Arms: Cellegesic (nitroglycerin 0.4%)
Drug: Placebo — Placebo was supplied as an ointment identical to Cellegesic ointment except that it contained no nitroglycerin.
  Arms: Placebo 375 mg

SUMMARY:
Anal fissure is a solitary ulcer in the squamous epithelium of the anus causing intense anal pain especially during defecation and for 1 or 2 hours afterwards. There are no approved drugs in the United States (US) for this condition and surgery is often the treatment choice. Strakan is conducting this confirmatory study so the product can be submitted for regulatory approval in the US. Strakan currently markets this product throughout Europe.

The objective of this study is to determine the effect of nitroglycerin ointment 0.4% (Cellegesic) versus placebo on average pain intensity over every 24 hour period for up to 21 days of treatment in 250 patients.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients of either sex.
* Between 18 and 75 years of age.
* With a single, chronic, posterior midline anal fissure.
* Defined as having anal pain for the 6 weeks prior to Screening.

Exclusion Criteria:

* More than one anal fissure.
* A fistula-in-ano or anal abscess.
* Inflammatory bowel disease.
* Fibrotic anal stenosis.
* Anal fissure secondary to an underlying condition.
* Any anal surgery.
* Concomitant medication that may interfere with study evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Clark, Study Director — Strakan Pharmaceuticals, Inc.

REFERENCES:
- [Derived] Berry SM, Barish CF, Bhandari R, Clark G, Collins GV, Howell J, Pappas JE, Riff DS, Safdi M, Yellowlees A. Nitroglycerin 0.4% ointment vs placebo in the treatment of pain resulting from chronic anal fissure: a randomized, double-blind, placebo-controlled study. BMC Gastroenterol. 2013 Jul 1;13:106. doi: 10.1186/1471-230X-13-106. PMID 23815124

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants applied placebo 375 mg ointment anally twice daily for 21 days. In addition, participants took acetaminophen 650 mg orally twice daily for 21 days.
Period: Overall Study
Arm/Group | Cellegesic (Nitroglycerin 0.4%) | Placebo
Started | 123 | 125
Received Treatment | 123 | 124
Completed | 106 | 113
Not Completed | 17 | 12
Not completed — Adverse Event | 9 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 4
Not completed — Voluntary withdrawal | 5 | 4
Not completed — Did not receive treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least 1 application of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cellegesic (Nitroglycerin 0.4%) | Placebo | Total
Number analyzed (Participants) | 123 | 124 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 114 | 117 | 231
  >=65 years | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.61) | 43.4 (13.22) | 45.0 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 116
  Male | 65 | 66 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 31 | 54
  Not Hispanic or Latino | 100 | 93 | 193
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 21 | 16 | 37
  White | 99 | 96 | 195
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Intensity at Days 14-18
Description: Participants rated the pain associated with their chronic anal fissure over the preceding 24 hours on a 100 mm visual analog scale at Baseline and on Days 14 through 18. The average pain rating on Days 14 through 18 was calculated and used to determine the change from Baseline. The left-end of the visual analog scale was labelled "least possible pain" and the right-end of the visual analog scale was labelled "worst possible pain". The pain rating ranged from 0 to 100, with a higher score indicating more pain. A negative change score indicated improvement.
Time Frame: Baseline to Day 18
Population: Intent-to-treat population: All randomized participants who had applied the study medication at least once.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Cellegesic (Nitroglycerin 0.4%) | Placebo
Number analyzed (Participants) | 123 | 124
Units on a scale | -40.4 (3.12) | -34.9 (3.04)

2. Secondary Outcome: Time to an Improvement in Pain Intensity
Description: Participants rated the pain associated with their chronic anal fissure over the preceding 24 hours on a 100 mm visual analog scale (VAS) at Baseline and on each of the 21 treatment days of the study. The left-end of the visual analog scale was labelled "least possible pain" and the right-end of the visual analog scale was labelled "worst possible pain". The pain rating ranged from 0 to 100, with a higher score indicating more pain. Improvement was defined as either a ≥ 50% decrease or a ≥ 10 mm decrease from Baseline in rated pain intensity.
Time Frame: Baseline to Day 21
Population: Intent-to-treat population: All randomized participants who had applied the study medication at least once. Only participants with an improvement in pain intensity were included in the analysis.
Measure: Mean (Standard Error); unit: Days
Groups:
- Cellegisic (Nitroglycerin 0.4%): Participants applied Cellegesic 375 mg ointment containing approximately 1.5 mg of nitroglycerin anally twice daily for 21 days. In addition, participants took acetaminophen 650 mg orally twice daily for 21 days.
Arm/Group | Cellegisic (Nitroglycerin 0.4%) | Placebo
Number analyzed (Participants) | 123 | 124
Days
  ≥ 50% decrease | 10.7 (0.6) | 13.2 (0.7)
  ≥ 10 mm decrease | 6.1 (0.5) | 7.2 (0.6)

3. Secondary Outcome: Percentage of Responders
Description: Participants rated the pain associated with their chronic anal fissure over the preceding 24 hours on a 100 mm visual analog scale at Baseline and on Days 14 through 18. The average pain rating on Days 14 through 18 was calculated. The left-end of the visual analog scale was labelled "least possible pain" and the right-end of the visual analog scale was labelled "worst possible pain". The pain rating ranged from 0 to 100, with a higher score indicating more pain. A responder was defined as a participant with either a ≥ 50% decrease or a ≥ 10 mm decrease from Baseline in the 24 hour average pain intensity averaged over Days 14 to 18.
Time Frame: Baseline to Day 18
Population: Intent-to-treat population: All randomized participants who had applied the study medication at least once.
Measure: Number; unit: Percentage of responders
Arm/Group | Cellegisic (Nitroglycerin 0.4%) | Placebo
Number analyzed (Participants) | 123 | 124
Percentage of responders
  ≥ 50% decrease | 72.4 | 64.5
  ≥ 10 mm decrease | 88.6 | 85.5

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 application of study medication.
Arm/Group | Cellegesic (Nitroglycerin 0.4%) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/123 | 1/124
Other Adverse Events (participants affected / at risk) | 96/123 | 67/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cellegesic (Nitroglycerin 0.4%) (N=123) | Placebo (N=124)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Anal sphincterotomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cellegesic (Nitroglycerin 0.4%) (N=123) | Placebo (N=124)
Headache (Nervous system disorders) | 86 | 59
Dizziness (Nervous system disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Sinusitis (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication statement in clinical trial agreement.